CLINICAL TRIAL: NCT05538169
Title: The Management of Radiotherapy-induced Hyposalivation Using Low-level Laser Therapy: A Case Series.
Brief Title: The Management of RT-induced Hyposalivation Using LLLT
Acronym: REACH-LLLT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: King Saud University (Other)
Responsible Party: Principal Investigator, Dr. Abdullah Mohamed Alsoghier, Assistant Professor of Oral Medicine, King Saud University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KingSaudU-E-21-6045
Record Dates: First submitted 2022-09-08; First posted 2022-09-13 (Actual); Last update posted 2023-10-23 (Actual); Status verified 2023-10

CONDITIONS: Head and Neck Cancer
MeSH Terms: conditions — Head and Neck Neoplasms

STUDY DESIGN:
Intervention Model Description: A prospective case series of patients who have received radiotherapy for SCC of the head and neck
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Laser therapy group (Experimental): There will be 2 weekly applications of a low-level laser diode (Pioon Laser) for a 4-week active treatment period. Thus, a total of 8 therapeutic sessions will be conducted
  Interventions: Device: low-level laser diode (Pioon Laser)

INTERVENTIONS:
Device: low-level laser diode (Pioon Laser) — Settings: the spot tip area of this tool is 0.088 cm2, semi-conductor diode, with a wavelength of 980 nm (near infrared), 200 mW output power, 1.97W/cm2 of power density, 3 J energy per point and application time 15 seconds per point].
  * PBM will apply punctually, in continuous emissions.
  * Extra-oral points: six points on each parotid gland, three points on each submandibular gland.
  * Intra-oral points: two points on each sublingual gland.
  * A total of 22 points will be applied in each session.

SUMMARY:
The primary purpose is to evaluate the effectiveness of photobiomodulation laser application in the management of patients with radiotherapy-induced hyposalivation. Secondary, to assess the changes in the scores of the patient's oral health-related quality of life using validated measurements.

DETAILED DESCRIPTION:
Head and neck cancer is a general term used to describe epithelial malignancies in the oral cavity, paranasal sinuses, nasal cavity, pharynx, and larynx. These malignancies are often presented as squamous cell carcinoma (SCC) of the head and neck with tobacco and alcohol consumption remaining the two main risk factors. In addition, human papillomavirus has been identified as another risk factor in a limited subset of these malignancies. More specifically, oral cancer accounts for 2%-4% of all cancer worldwide with 90% of these cases presented as SSC worldwide compared to 44.8% in Saudi Arabia. Clinically, patients often presented with white and/or red patches, hoarseness, non-healed ulcers, throat pain, and painless cervical lump which may persist for more than 3 weeks period.

Most head & neck cancer patients who received radiotherapy are likely to experience xerostomia and salivary glands hypofunction, mucositis, and possibly the loss of taste.

Furthermore, the effect of hyposalivation is not only limited to taste dysfunction but also associated with opportunistic infections, difficulty in chewing and speaking, rapid progression of caries, and oral mucositis. All these secondary complications are usually associated with pain and discomfort which will heavily affect the patient quality of life if they are untreated. Treatment options include moisturizing agents or artificial saliva which have a palliative effect however they are not preferred nor accepted by most patients.

The outcome of low-level laser therapy usage on cancer patients is well documented and well established in the literature. The vast majority of the results suggest that this therapy is an effective treatment option to stimulate salivary glands flow and decrease xerostomia/hyposalivation symptoms. In the present study, the efficiency of this treatment option will be tested as well as the changes in the patient's quality of life during and after the radiation treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 and above
* Clinically diagnosed with hyposalivation [an unstimulated salivary flow rate of ≤ 0.1ml per minute] (31) due to recent radiation therapy of SCC of the head and neck.

Exclusion Criteria:

* Individuals with systemic diseases that could affect the salivary glands function such as (e.g. Sjogren syndrome) and medications (e.g. beta-blockers and diuretics for hypertension).
* Individuals who had an allergy to toluidine blue stain.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2022-01-03 (Actual); Primary Completion 2023-08-01 (Actual); Study Completion 2023-10-01 (Actual)

PRIMARY OUTCOMES:
Unstimulated and stimulated salivary flow rate | 12 weeks
  The unstimulated and stimulated salivary flow rate (ml/minute) will be collected at three different time periods: (T1) the first visit and before applying the laser, (T2) the 8th visit and after using the laser, and (T3) the re-evaluation visit after two months.

SECONDARY OUTCOMES:
Xerostomia assessment | 12 weeks
  Xerostomia will be analysed at (T1) first visit, (T2) 8th visit, and (T3) at the re-evaluation visit using the Arabic version of Xerostomia Inventory, which is assessed by a 4-point scale (from never = 0 to always = 3).
Dysgeusia assessment | 12 weeks
  Dysgeusia will be analysed at (T1) first visit, (T2) 8th visit, and (T3) at the re-evaluation visit using the 11-item Dysguesia Questionnaire, which is assessed by a mix of choices (e.g. yes or no) and 4-point scale for each question (little, tolerably, a lot or don't rememeber).
Quality of life assessment | 12 weeks
  The Oral health-related quality of life (OHQoL) will be measured at (T1) first visit, (T2) 8th visit, and (T3) at the re-evaluation visit using the validated Arabic version of Oral Health Impact Profile (OHIP-5), which is which is assessed by a 5-point scale (from never = 0 to always = 4).

CONTACTS AND LOCATIONS:
Locations (1):
- King Saud Universiry, Riyadh, Saudi Arabia

REFERENCES:
- [Derived] Alsoghier A, Mutaieb S, Bukhari A, AlQarni M, Alhazzaa S, Aljabab S, Alsuhaibani A, Faden A. Management of radiotherapy-induced hyposalivation using photobiomodulation therapy: a case series. Lasers Med Sci. 2025 Jan 20;40(1):25. doi: 10.1007/s10103-025-04292-3. PMID 39833441